CLINICAL TRIAL: NCT05242822
Title: A Phase 1/1b, Open-label, Multicenter Study to Investigate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Anti-tumor Activity of KIN-3248 in Participants With Advanced Tumors Harboring FGFR2 and/or FGFR3 Gene Alterations
Brief Title: A Study to Evaluate KIN-3248 in Participants With Advanced Tumors Harboring FGFR2 and//or FGFR3 Gene Alterations
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to a change in the Sponsor's corporate strategy the study was terminated early by the Sponsor prior to enrollment into the dose expansion part of the study (Part B).
Sponsor: Kinnate Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KN-4802
Record Dates: First submitted 2022-01-26; First posted 2022-02-16 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2024-12

CONDITIONS: Solid Tumor, Adult; Intrahepatic Cholangiocarcinoma; Urothelial Carcinoma
Keywords: FGFR inhibitor; targeted therapy; FGFR2 alteration; FGFR3 alteration; secondary resistance; FGFR alteration
MeSH Terms: conditions — Cholangiocarcinoma; Carcinoma, Transitional Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part A - dose escalation (Experimental): Dose escalation of KIN-3248 in patients with solid tumors
  Interventions: Drug: KIN-3248
- Part B - dose expansion (Experimental): Dose expansion evaluating the recommended dose and schedule of KIN-3248 identified from Part A
  Interventions: Drug: KIN-3248

INTERVENTIONS:
Drug: KIN-3248 — KIN-3248 will be administered orally once daily in 28-day cycles

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics (PK), and preliminary efficacy of KIN-3248, an oral small molecule FGFR inhibitor, in adults with advanced tumors harboring FGFR2 and/or FGFR3 gene alterations.

DETAILED DESCRIPTION:
This is a two-part, open label, multi-center, dose escalation and dose expansion study in participants with advanced tumors harboring FGFR2 and/or FGFR3 gene alterations.

Part A (dose escalation) is aimed at evaluating the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of KIN-3248, and determining the maximum tolerated dose (MTD) of daily dosing of KIN-3248.

Part B (dose expansion) may open once either the MTD and/or a biologically active dose of KIN-3248 is identified. Part B is aimed at evaluating the safety and efficacy of KIN-3248 at the recommended dose and schedule in participants with cancers harboring FGFR2 and/or FGFR3 gene alterations, including intrahepatic cholangiocarcinoma (ICC), urothelial cancer (UC), and other solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent prior to initiation of any study-specific procedures
* Advanced stage solid tumor
* Known FGFR2 and/or FGFR3 gene alteration, as confirmed by previous genomic analysis of tumor tissue or ctDNA
* Measurable or evaluable disease according to RECIST v1.1
* ECOG performance status 0 or 1
* Adequate organ function, as measured by laboratory values (criteria listed in protocol)
* Able to swallow, retain, and absorb oral medications

Exclusion Criteria:

* Known clinically-active or clinically-progressive brain metastases from non-brain tumors
* History and/or current evidence of abnormal calcium-phosphorous homeostasis, ectopic mineralization or calcification, or corneal or retinal disorder/keratopathy
* GI tract disease causing an inability to take oral medication, malabsorption syndrome, requirement for intravenous alimentation, or uncontrolled inflammatory GI disease
* Active, uncontrolled bacterial, fungal, or viral infection
* Women who are lactating or breastfeeding, or pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2022-03-29 (Actual); Primary Completion 2024-10-03 (Actual); Study Completion 2024-10-03 (Actual)

PRIMARY OUTCOMES:
Part A (dose escalation) - incidence of dose limiting toxicities (DLTs) | Initiation of study drug through 28 days
Part A (dose escalation) - incidence of adverse events (AEs) | Initiation of study drug through 28 days after last dose (up to approximately 18 months)
Part B (dose expansion) - objective response rate (ORR): the proportion of participants who have achieved partial response (PR) or complete response (CR) according to RECIST v1.1 | Initiation of study drug until disease progression (up to approximately 36 months)
Part B (dose expansion) - disease control rate (DCR): the proportion of participants who achieve stable disease, PR, or CR | Initiation of study drug until disease progression (up to approximately 36 months)
Part B (dose expansion) - duration of response (DOR): the length of time between initial tumor response to documented tumor progression | Initiation of study drug until disease progression (up to approximately 36 months)
Part B (dose expansion) - progression-free survival (PFS): the length of time until documented tumor progression | Initiation of study drug until disease progression (up to approximately 36 months)

SECONDARY OUTCOMES:
Part A (dose escalation) - PK - maximum plasma concentration (Cmax) of KIN-3248 | Initiation of study drug through Cycle 5 (up to approximately 4 months)
Part A (dose escalation) - PK - time to reach maximum plasma concentration (Tmax) of KIN-3248 | Initiation of study drug through Cycle 5 (up to approximately 4 months)
Part A (dose escalation) - PK - area under the plasma concentration-time curve (AUC) of KIN-3248 | Initiation of study drug through Cycle 5 (up to approximately 4 months)

CONTACTS AND LOCATIONS:
Locations (21):
- United States (12):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Mayo Clinic Florida, Jacksonville, Florida
  - Sarah Cannon Research Institute - Lake Nona, Orlando, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - START Midwest, Grand Rapids, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - NYU Langone Cancer Center, New York, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
- Beijing Cancer Hospital, Beijing, Haidian District, China
- Rigshospitalet (Copenhagen University Hospital) - Finsencentret - Onkologisk Klinik, Copenhagen, Denmark
- South Korea (3):
  - Seoul National University Hospital (SNUH), Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
- START (Fundacion Jimenez Diaz), Madrid, Madrid, Spain
- Taiwan (3):
  - National Taiwan University Hospital, Taipei, Taiwan
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - Veterans General Hospital - Taipei, Taipei